CLINICAL TRIAL: NCT01841671
Title: A Phase 4, Randomized, Open-Label Study to Assess Humoral and Intestinal Polio Immunity Following a Three-Dose Trivalent Inactivated Polio Vaccine Schedule Relative to Two Sequential Schedules of IPV/Bivalent Oral Polio Vaccines
Brief Title: Immunogenicity of 1 or 2 Doses of bOPV in Chilean Infants Primed With IPV Vaccine
Acronym: IPV002ABMG
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chile (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, Miguel O'Ryan Gallardo, Full Professor and Associate Director for Innovation, Faculty of Medicine, University of Chile, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPV002ABMG
Record Dates: First submitted 2013-04-19; First posted 2013-04-26 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-04

CONDITIONS: Polio
Keywords: Polio; IPV; bOPV; mOPV; vaccination
MeSH Terms: conditions — Poliomyelitis | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IPV/IPV/IPV/Rotarix/mOPV type 2 (Experimental): 190 healthy infants due for their first dose of polio vaccines will be receive IPV, IPV, IPV at 8, 16 and 24 weeks of age respectively, Rotarix at 8 and 16 weeks if parents accept (optional), and mOPV type 2 at 28 weeks of age
  Interventions: Biological: IPV; Biological: mOPV type 2; Biological: Rotarix
- IPV/IPV/bOPV/Rotarix/mOPV type 2 (Active Comparator): 190 healthy infants due for their first dose of polio vaccines will be receive IPV, IPV, bOPV at 8, 16 and 24 weeks of age respectively and Rotarix at 8 and 16 weeks f age (optional) and mOPV type 2 at 28 weeks of age
  Interventions: Biological: IPV; Biological: bOPV; Biological: mOPV type 2; Biological: Rotarix
- IPV/bOPV/bOPV/Rotarix/mOPV type 2 (Active Comparator): 190 healthy infants due for their first dose of polio vaccines will be receive IPV, bOPV, bOPV at 8, 16 and 24 weeks of age respectively and Rotarix at 8 and 16 weeks of age (optional)and mOPV type 2 at 28 weeks of age
  Interventions: Biological: IPV; Biological: bOPV; Biological: mOPV type 2; Biological: Rotarix

INTERVENTIONS:
Biological: IPV — Blood samples for poliovirus neutralizing antibodies to be obtained as follows: Group 1 at weeks 8, 16, 28 and 29; Group 2 and 3 at 8, 24, 28 and 29. Stool samples for poliovirus cuantification, for all groups, to be obtained at weeks 28, 29, 30, 31, 32.
  Other Names: Sanofi IPV
Biological: bOPV — As indicated
  Other Names: Sanofi bOPV
  Arms: IPV/IPV/bOPV/Rotarix/mOPV type 2; IPV/bOPV/bOPV/Rotarix/mOPV type 2
Biological: mOPV type 2 — Administered at 28 weeks of age to all study participants
  Other Names: GSK mOPV type 2
Biological: Rotarix — Administered at 8 and 16 weeks to all study participants accepting to recive this vaccine
  Other Names: GSK Rotarix

SUMMARY:
The rationale for this study (IPV 002ABMG) is to evaluate and compare three doses of IPV, two doses of IPV plus one bOPV, and one dose of IPV plus two doses of bOPV in order to provide evidence for better immunization policy making in regions of the world that must switch to use of IPV/bOPV schedules in the 2014-2015 time frame. The goal is to identify the best option optimizing humoral immune responses, intestinal immunity and thereby prevent community transmission as well as preventing VAPP. Specifically, the study seeks to show that both of the sequential regimens are equivalent (not-inferior) to the 3-dose IPV regimen in the seroconversion rates to both type 1 and type 3 poliovirus such that not more than 10% of subjects fall below the 95% confidence interval observed for the 3-dose IPV alone regimen and the geometric mean titers (GMTs) are no more than 2/3 logs less than those for the 3-dose IPV regimen. In addition, the study will evaluate by a novel method (poliovirus shedding index), the adequacy of IPV vaccines in inducing intestinal immunity, specifically by reducing the shedding of poliovirus type 2 after an OPV challenge. The hypotheses of the study are:

* A 3-dose IPV/bOPV sequential schedule including 1 or 2 doses of bOPV is non-inferior in terms of types 1 and 3 seroconversion rates and GMTs to a 3-dose IPV schedule.
* Two and possibly 1 IPV dose(s) provides significant seroconversion rates and GMTs to type 2 poliovirus and sufficient priming to induce a rapid immune response in the context of an oral challenge at 7 months of age.
* Three, 2, and possibly 1 dose of IPV will induce intestinal immunity to poliovirus type 2 as measured by a combination of quantity of virus in stools and duration of shedding (shedding index).

In addition to these 3 hypotheses, the study will explore the following hypothesis:

• Co-administration of bOPV and rotavirus at 16 weeks of age (the second rotavirus dose) provides similar antirotavirus IgA seroconversion rates and GMCs compared to subjects receiving rotavirus vaccine together with IPV.

DETAILED DESCRIPTION:
3.0 STUDY DESIGN This is a multicenter, randomized, unblinded study. Healthy infants attending the well-child care at outpatient clinics and due for their first dose of polio vaccines will be eligible for the study. Infants 8 wks ± 7 days of age will be randomized and allocated to three treatment groups.

4.0 STUDY POPULATION The study will be conducted in up to 7 "vacunatorios" in Chile. Parents or legal guardians of healthy infants, who are receiving well-child care at designated outpatient clinics, will be approached to participate in the study.

5.0 TREATMENT OF SUBJECTS 5.1 Vaccines The vaccines to be used in this study include bOPV, mOPV2, and IPV (see Section 14.2 for package inserts).

5.1.1 Bivalent Oral Polio Vaccine (bOPV) Produced by Sanofi Pasteur, Lyon, France, bivalent OPV vaccine contains types 1 and 3 polioviruses and it is indicated for supplementary immunization activities in children from 0 to 5 years of age to prevent or contain outbreaks caused by these 2 serotypes. The vaccine contains at least 6.0 log CCID50 of LS c2ab live attenuated polio virus type 1; and at least 5.8 log CCID50 Leon I2aIb strain of polio virus type 3. The vaccine dose is 2 drops (0.1 mL) using a multi-dose dropper vial, given directly into the mouth. The vaccine should be stored in a freezer at -20°C, and after thawing it can be stored up to 6 months at refrigerated temperatures of +2 to +8°C.

5.1.2 Monovalent Oral Polio Vaccine Type 2 (mOPV2) Monovalent OPV type 2 live attenuated poliomyelitis virus vaccine (mOPV2) is produced by Glaxo SmithKline, Rixensart, Belgium, as a sterile suspension of poliovirus serotype 2 for oral administration. Each dose (0.1 mL) contains not less than 105.0 CCID50 of the Sabin strain type 2 (P 712, Ch, 2ab). This will be the challenge OPV strain used to assess intestinal shedding and immunity. The vaccine should be stored in a freezer at -20°C, and after thawing it can be stored up to 6 months at refrigerated temperatures of +2 to +8°C.

5.1.3 Inactivated Polio Vaccine (IPV) Inactivated poliovirus vaccine is produced by Sanofi-Pasteur as a sterile suspension of 3 types of poliovirus. Each dose of vaccine (0.5 mL) contains 40 D antigen units of Mahoney strain (Type 1); 8 D antigen units of MEF-1 strain (Type 2); and 32 D antigen units of Saukett strain (Type 3). It also contains 0.5% of 2-phenoxyethanol and a maximum of 0.02% of formaldehyde as preservatives. It may also contain 5 ng of neomycin, 200 ng of streptomycin, and 25 ng of polymixin B as residuals of the vaccine production. The vaccine does not contain Thimerosal. The vaccine should be kept refrigerated at +2 to +8°C, and should never be frozen. The dose of IPV vaccine should be 0.5 mL administered intramuscularly in the anterolateral aspect of the thigh.

5.2 Vaccine Intervals and Administration All polio vaccine doses should be administered at least 4 weeks or more apart. For IPV, the administration site is restricted to the anterolateral aspect of the left thigh.

* All other intramuscular (IM) EPI routine vaccines will be administered to the anterolateral aspect of the right thigh (or the arm at 16 weeks when 3 vaccines are to be administered including IPV, pentavalent combination vaccine, and S. pneumoniae). These vaccines should not be injected in the gluteal area or areas where there may be a major nerve damage.
* IPV will be administered IM at Week 8 (Group 1), Weeks 8 and 16 (Group 2), or Weeks 8, 16, and 24 (Group 3).
* Bivalent OPV will be administered as oral drops (2 drops for each vaccination) at Weeks 16 and 24 (Group 1) or Week 24 (Group 2).
* An oral challenge dose (2 drops) of mOPV2 will be administered at Week 28.

Prior to an injection of any vaccine, all known precautions should be taken to prevent adverse reactions. This includes a review of the potential participant's history with respect to possible allergic reactions to the vaccine or similar vaccines. Epinephrine Injection (1:1000) and other appropriate agents should be available to control immediate allergic reactions. Health-care providers should obtain the previous immunization history of the subject, and inquire about the current health status of the subject.

Infants participating in the study will be provided the recommended vaccines aside from polio vaccine as per the National Immunization Schedule of Chile (DTPw/HBV/Hib, S. pneumoniae vaccine).

In addition, a 2-dose (RotarixTM) oral rotavirus vaccine will be offered during the study at 8 weeks and 16 weeks of age.

Serology Testing

Rational for each blood sample: After thorough discussions on the minimum number of serum samples required to obtain valid answers to our hypothesis, the research group has arrived to the following:

1. Baseline serum sample at 7-8 weeks to determine antibody titers to polioviruses (and rotavirus) before any vaccination, required as a basis to detect seroconversion rates.
2. Post IPV dose 1 at 16 weeks (Group 1) or IPV 2 at 24 weeks (Groups 2 and 3) to determine IPV/bOPV dose-dependent seroconversions for poliovirus 2 with the shortest possible latency after vaccination to avoid the potential confounder associated with exposure to circulating poliovirus 2 vaccine viruses.
3. Post 3 doses to measure the primary objective, seroconversion and GMTs to types 1 and 3 after the different schedules. This serum will also be used for antirotavirus antibody determinations in order to calculate seroconversion rates and GMCs achieved.
4. One week post-type 2 live poliovirus vaccine challenge at 28 weeks to determine if infants who have not seroconverted to type 2 poliovirus after completing the series of 3 immunizations at 8, 16, and 24 weeks in each of the 3 groups, do so rapidly within 1 week after the challenge. Seroconversion within 1 week strongly suggests that although the individual had not seroconverted prior to the mOPV2 challenge, that they would do so rapidly should they encounter cVDPV2 in the environment; this in turn suggests that although they might become infected by cVDPV2, their risk of developing neuroparalytic disease as a consequence would nonetheless be substantially reduced.

A total of 4 blood samples will be collected for each study subject. A maximum of 3 mL will be obtained by heel stick or venipuncture methods. Each blood sample will be transported within 24 hours in appropriate cold chain conditions to the "Central Study Laboratory" at the Microbiology and Mycology Program, Institute of Biomedical Sciences, Faculty of Medicine, University of Chile. Sera will be obtained and 2 aliquots will be placed into cryovials, labeled with linked coding, and stored in a -20°C freezer. One aliquot will be shipped in appropriate cold chain conditions to the Polio and Picornavirus Laboratory Branch, Center for Disease Control and Prevention. The second aliquot will be left on repository storage at the study center.

Sera will be processed following a standard protocol (see Section 14.1). Neutralizing antibodies against polioviruses 1, 2, and 3 will be determined using a sero-neutralization assay. The laboratory will be blinded with regard to the vaccination status of individuals contributing particular specimens, ensuring the integrity of the study. After successful completion of testing, duplicate specimens will be destroyed. Authorized specimens assays are only for antibody levels to valences included in the study vaccines. Should the case arise, the use of these specimens for any other assay will require the approval of the study Sponsor and the Principal Investigator, as well as Institutional Review Board (IRB) or Independent Ethics Committee (IEC) approval, as per applicable rules and regulations.

Baseline sera and sera obtained at 28 weeks will be processed for antirotavirus IgA concentration as previously described at Glaxo SmithKline laboratories (26).

5.3 Stool Samples for Poliovirus "Shedding Index" determination Stool samples (5 to 10 grams) will be collected at 5 times for each subject, using WHO approved protocols and kits, and transported and stored following the WHO procedures for detection of polioviruses. Fresh stools will be collected unmixed with urine in a screw-top container, placed in a cold box with frozen ice packs, and transported to the designated laboratory for storage in a freezer at -20°C. A log book of collected and stored samples will be kept by the study personnel. Stool samples will be used later to determine the excretion of polioviruses as per protocol (Section 14.1). Samples will be sent in batches to the reference laboratory for poliovirus culture.

5.4 Medications/Treatments Permitted (including rescue medication) and not Permitted Before and/or During the Trial There will be no restrictions in using medications/treatments except for the following conditions: primary immune deficiency or immune deficiency subsequent to treatment, leukemia, lymphoma or advanced malignancy in the subject to be vaccinated or his/her close contact. Only medications to treat SAEs or IMEs will be documented in eCRF. All other medications will be captured and recorded in the source document at the investigators discretion at the investigational site.

5.5 Subject Compliance Subjects are required to abide by scheduled visits and the vaccine schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 8 weeks (-7 to +7 days).
2. Healthy infants of all ethnicities and both genders without obvious medical conditions that preclude the subject to be in the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 parent or legal guardian who, in the opinion of the investigator, is capable of understanding and complying with the protocol requirements.

Exclusion Criteria:

1. Previous vaccination against poliovirus.
2. Low birth weight (BW <2,500 grams).
3. Twins or multiple pregnancy infants.
4. Another family or household member who has received OPV within the past 6 months or is going to receive OPV within the following 6 months.
5. Any confirmed or suspected immunosuppressive or immunedeficient condition including human immunodeficiency virus (HIV) infection.
6. Family history of congenital or hereditary immunodeficiency.
7. Major congenital defects or serious chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
8. Known allergy to any component of the study vaccines.
9. Uncontrolled coagulopathy or blood disorder contraindicating intramuscular injections.
10. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
11. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 7 Weeks to 9 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 570 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Types 1 and 3 poliovirus humoral immune response | 12 months
  Two primary endpoints will be used as the basis for evaluation of the IPV/OPVb sequential regimens compared to three doses of IPV:
  * Seroconversion to type 1 (type-specific titers ≥1:8 and > 4-fold over expected levels of maternally-derived antibody) and GMTs achieved at 28 weeks.
  * Seroconversion to type 3 (type-specific titers ≥1:8 and > 4-fold over expected levels of maternally-derived antibody) and GMTs achieved at 28 weeks.

SECONDARY OUTCOMES:
Poliovirus Type 2 humoral and intestinal immune response and safety | 12 months (18 months for intestinal immunity)
  * Seroconversion to type 2 (type-specific titers ≥1:8 and > 4-fold over expected levels of maternally-derived antibody) and GMTs achieved after 1 dose of IPV at 16 weeks, after 2 doses at 24 weeks, after 3 doses at 28 weeks, and after the mOPV type 2 challenge dose at 29 weeks.
  * Viral shedding index for type 2 virus following mOPV2 challenge (28-day area under the curve [AUC] of quantitative virus shedding at Days 7, 14, and 21 post-mOPV2 challenge).
  * Safety Endpoints: SAEs as defined in the protocol throughout the study period and IMEs as defined in the protocol up to 28 days post-vaccination.

OTHER OUTCOMES:
antirotavirus IgA seroconversion rates | 18 months
  • Antirotavirus IgA seroconversion (> 20 units/mL) and GMCs after the second dose of RotarixTM at 16 weeks of age.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L O'Ryan, MD, Principal Investigator — University of Chile
Locations (1):
- Facultad de Medicina de la Universidad de Chile, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] 1. Global Polio Eradication Initiative. Data and Monitoring: Polio this week. Available at http://www.polioeradication.org/Dataandmonitoring/Poliothisweek.aspx.http://www.polioeradication.org/Dataandmonitoring/Poliothisweek.aspx. Copyright 2010. Accessed 8/23/2012 2. Sixty-fifth World Health Assembly. Poliomyelitis: Intensification of the global eradication initiative. WHA 65.5, Agenda item 13.10; 26 May 2012. 3. Sabin, A B.
- [Background] 2. Sixty-fifth World Health Assembly. Poliomyelitis: Intensification of the global eradication initiative. WHA 65.5, Agenda item 13.10; 26 May 2012.
- [Background] Asturias EJ, Dueger EL, Omer SB, Melville A, Nates SV, Laassri M, Chumakov K, Halsey NA. Randomized trial of inactivated and live polio vaccine schedules in Guatemalan infants. J Infect Dis. 2007 Sep 1;196(5):692-8. doi: 10.1086/520546. Epub 2007 Jul 23. PMID 17674310
- [Background] Minor PD. Polio eradication, cessation of vaccination and re-emergence of disease. Nat Rev Microbiol. 2004 Jun;2(6):473-82. doi: 10.1038/nrmicro906. No abstract available. PMID 15152203
- [Derived] Brickley EB, Wieland-Alter W, Connor RI, Ackerman ME, Boesch AW, Arita M, Weldon WC, O'Ryan MG, Bandyopadhyay AS, Wright PF. Intestinal Immunity to Poliovirus Following Sequential Trivalent Inactivated Polio Vaccine/Bivalent Oral Polio Vaccine and Trivalent Inactivated Polio Vaccine-only Immunization Schedules: Analysis of an Open-label, Randomized, Controlled Trial in Chilean Infants. Clin Infect Dis. 2018 Oct 30;67(suppl_1):S42-S50. doi: 10.1093/cid/ciy603. PMID 30376086
- [Derived] O'Ryan M, Bandyopadhyay AS, Villena R, Espinoza M, Novoa J, Weldon WC, Oberste MS, Self S, Borate BR, Asturias EJ, Clemens R, Orenstein W, Jimeno J, Ruttimann R, Costa Clemens SA; Chilean IPV/bOPV study group. Inactivated poliovirus vaccine given alone or in a sequential schedule with bivalent oral poliovirus vaccine in Chilean infants: a randomised, controlled, open-label, phase 4, non-inferiority study. Lancet Infect Dis. 2015 Nov;15(11):1273-82. doi: 10.1016/S1473-3099(15)00219-4. Epub 2015 Aug 26. PMID 26318714